CLINICAL TRIAL: NCT02306057
Title: Interstitial Colloid Osmotic Pressure in Children With Congenital Heart Defect Preparing for Fontan Surgery Undergoing Preoperative Catheterization and Surgery in General Anesthesia
Brief Title: Fluid Balance in Children Undergoing Fontan Surgery
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Marianne Indrebo, MD Research fellow, Oslo University Hospital
Other Study IDs: 063.09b
Record Dates: First submitted 2014-10-31; First posted 2014-12-03 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Heart Defects, Congenital; Hypoplastic Left Heart Syndrome
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Interstitial fluid Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pre BCPC: Children undergoing catheterization before Bidirectional CavoPulmonary Connection (BCPC) procedure
  Interventions: Procedure: Pre BCPC
- BCPC surgery: Children undergoing surgical BCPC procedure
  Interventions: Procedure: BCPC surgery
- Pre TCPC: Children undergoing catheterization before Total CavoPulmonary Connection (TCPC )procedure
  Interventions: Procedure: Pre TCPC
- TCPC surgery: Children undergoing surgical TCPC procedure
  Interventions: Procedure: TCPC

INTERVENTIONS:
Procedure: Pre BCPC — Routine catheterization before surgical procedure Bidirectional CavoPulmonary Connection
  Groups: Pre BCPC
Procedure: Pre TCPC — Routine catheterization before surgical procedure Total CavoPulmonary Connection
  Groups: Pre TCPC
Procedure: BCPC surgery — Surgical procedure Bidirectional CavoPulmonary Connection
  Groups: BCPC surgery
Procedure: TCPC — Surgical procedure Total CavoPulmonary Connection
  Groups: TCPC surgery

SUMMARY:
This project will evaluate fluid balance and edema formation in children with congenital heart disease in need of a surgical procedure, The Fontan procedure. Surgery will make the child end up with a univentricular heart with one-chamber circulation ( Fontan circulation). This project will evaluate if these children has increased micro vascular leakage before surgery due to their congenital heart defect. The project will also investigate if the edema formation seen during cardiac surgery with the use of Cardio-Pulmonary Bypass (CPB) and hypothermia is caused by capillary leakage of plasma protein.

The study hypothesis are

1. Edema developed during heart surgery is caused by reduced colloid osmotic pressure gradient through the capillary membrane.
2. The degree of micro vascular leakage in open-heart surgery is related to duration of CPB and hypothermia.
3. Fontan circulation cause peripheral edema related to elevated central venous pressure and is not caused by increased micro vascular leakage of plasma proteins.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of Congenital heart defect in need of Fontan procedure -

Exclusion Criteria: No parental consent

-

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with congenital heart defect scheduled for Fontan surgery
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-11; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Interstitial colloid osmotic pressure | Before and after surgery or catheterization
  Change in interstitial colloid osmotic pressure

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Indrebø, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Indrebo M, Berg A, Holmstrom H, Seem E, Guthe HJT, Wiig H, Norgard G. Fluid accumulation in the staged Fontan procedure: the impact of colloid osmotic pressures. Interact Cardiovasc Thorac Surg. 2019 Apr 1;28(4):510-517. doi: 10.1093/icvts/ivy298. PMID 30371784